CLINICAL TRIAL: NCT01179568
Title: Optimizing Treatment for Complicated Grief (Healing Emotions After Loss:HEAL)
Brief Title: A Study of Medication With or Without Psychotherapy for Complicated Grief
Acronym: HEAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5971; R01MH060783 (NIH)
Record Dates: First submitted 2010-07-14; First posted 2010-08-11 (Estimated); Results first posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-11

CONDITIONS: Complicated Grief; Bereavement
Keywords: Grief; Bereavement; Psychotherapy; Medication; Treatment study
MeSH Terms: interventions — Citalopram; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CGT with Citalopram (Active Comparator): Targeted psychotherapy for complicated grief will be combined with SSRI medication.
  Interventions: Drug: Citalopram; Behavioral: Complicated Grief Treatment
- Citalopram (Active Comparator): Citalopram is an Selective Serotonin Reuptake Inhibitor (SSRI) medication. It will be combined with grief-focused clinical management.
  Interventions: Drug: Citalopram
- Placebo (Sugar pill) (Placebo Comparator): Inactive medication. It will be combined with grief-focused clinical management.
  Interventions: Other: Placebo
- CGT with Placebo (Active Comparator): The targeted psychotherapy for complicated grief will be combined with inactive medication.
  Interventions: Behavioral: Complicated Grief Treatment; Other: Placebo

INTERVENTIONS:
Drug: Citalopram — 16 weeks of medication provided flexibly up to 40 mg/day. Medication will be administered in a double-blind fashion.
  Other Names: Celexa
  Arms: CGT with Citalopram; Citalopram
Behavioral: Complicated Grief Treatment — Complicated Grief Treatment (CGT) is a targeted psychotherapy for complicated grief. The treatment integrates principles, strategies and techniques from interpersonal psychotherapy, trauma-focused cognitive behavioral treatment and motivational interviewing. Treatment includes 16 sessions provided within 20 weeks.
  Other Names: CGT
  Arms: CGT with Citalopram; CGT with Placebo
Other: Placebo — 16 weeks of daily inactive medication. It will be administered in a double-blind fashion.
  Other Names: Sugar pill
  Arms: CGT with Placebo; Placebo (Sugar pill)

SUMMARY:
The major goal of this 4-site, double blind, placebo-controlled intervention trial is to assess the efficacy of medication (Citalopram) alone or with psychotherapy (Complicated Grief Therapy) to treat the symptoms of complicated grief.

DETAILED DESCRIPTION:
Complicated grief (CG) is a debilitating condition that is estimated to affect millions of people in the United States alone. We conducted the first randomized controlled study to address this condition (MH60783) and confirmed efficacy of a targeted psychotherapy, complicated grief treatment (CGT). Participants in our prior study continued stable antidepressant medication while receiving CGT or Interpersonal Psychotherapy (IPT). Individuals taking antidepressants had better outcome in both treatments, though CGT was superior to IPT when administered with (60% responders v. 40%) or without (42% v.19%) antidepressants. Studies of antidepressant medication alone have shown mixed results with SSRIs appearing to be promising. However, there has been no randomized controlled study of SSRIs for CG. Determining the efficacy of SSRI treatment for CG, when administered with and without CGT, is of great public health importance.

We assembled 4 groups of investigators with strong track records in bereavement research and extensive experience with intervention studies and multicenter projects, to conduct a study of citalopram (CIT) efficacy. We plan to enroll participants with a primary diagnosis of Complicated Grief and randomly assign them (n=480; 50 at Columbia) to receive treatment with CIT, Placebo (PBO), CIT + CGT or PBO + CGT over a period of approximately 16 weeks. We want to determine whether citalopram shows a better response than placebo, when administered either with or without CGT. We will also address the question of whether CIT performs as well when administered alone as it does when administered with CGT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Complicated Grief and this is the patient's most important (primary) problem
* Ability to give informed consent
* Fluent in English
* Willingness to have sessions audiotaped
* Willingness to undergo random assignment

Exclusion Criteria:

* Diagnosis of one or more of the following disorders: Schizophrenia or other psychotic disorder, current (past 6 months) substance abuse, Bipolar Disorder, current manic episode, Dementia
* Pregnant or lactating women and women of childbearing potential not using medically accepted forms of contraception
* Acute, unstable or severe medical illness such as (but not limited to) stroke, epilepsy, or other neurodegenerative disorders, metastatic or active cancer, hepatic disease, or primary renal disease requiring dialysis
* Prior intolerance of citalopram
* Pending or active disability claim or lawsuit related to the death

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2010-03; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Shear, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - VASDHS / University of California San Diego, San Diego, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York State Psychiatric Institute, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Simon NM, Thompson EH, Pollack MH, Shear MK. Complicated grief: a case series using escitalopram. Am J Psychiatry. 2007 Nov;164(11):1760-1. doi: 10.1176/appi.ajp.2007.07050800. No abstract available. PMID 17974946
- [Background] Shear K, Frank E, Houck PR, Reynolds CF 3rd. Treatment of complicated grief: a randomized controlled trial. JAMA. 2005 Jun 1;293(21):2601-8. doi: 10.1001/jama.293.21.2601. PMID 15928281
- [Background] Schwartz D, Lellouch J. Explanatory and pragmatic attitudes in therapeutical trials. J Chronic Dis. 1967 Aug;20(8):637-48. doi: 10.1016/0021-9681(67)90041-0. No abstract available. PMID 4860352
- [Background] Tunis SR, Stryer DB, Clancy CM. Practical clinical trials: increasing the value of clinical research for decision making in clinical and health policy. JAMA. 2003 Sep 24;290(12):1624-32. doi: 10.1001/jama.290.12.1624. PMID 14506122
- [Background] Jacobs SC, Nelson JC, Zisook S. Treating depressions of bereavement with antidepressants. A pilot study. Psychiatr Clin North Am. 1987 Sep;10(3):501-10. PMID 3684751
- [Background] Shear MK. Clinical practice. Complicated grief. N Engl J Med. 2015 Jan 8;372(2):153-60. doi: 10.1056/NEJMcp1315618. No abstract available. PMID 25564898
- [Derived] Calderon A, Irwin M, Simon NM, Shear MK, Mauro C, Zisook S, Reynolds CF 3rd, Malgaroli M. Depression is Associated with Treatment Response Trajectories in Adults with Prolonged Grief Disorder: A Machine Learning Analysis. medRxiv [Preprint]. 2024 Dec 12:2024.12.11.24318861. doi: 10.1101/2024.12.11.24318861. PMID 39711702
- [Derived] Na PJ, Adhikari S, Szuhany KL, Chen AZ, Suzuki RR, Malgaroli M, Robinaugh DJ, Bui E, Mauro C, Skritskaya NA, Lebowitz BD, Zisook S, Reynolds CF 3rd, Shear MK, Simon NM. Posttraumatic Distress Symptoms and Their Response to Treatment in Adults With Prolonged Grief Disorder. J Clin Psychiatry. 2021 Apr 20;82(3):20m13576. doi: 10.4088/JCP.20m13576. PMID 34000119
- [Derived] Zisook S, Shear MK, Reynolds CF, Simon NM, Mauro C, Skritskaya NA, Lebowitz B, Wang Y, Tal I, Glorioso D, Wetherell JL, Iglewicz A, Robinaugh D, Qiu X. Treatment of Complicated Grief in Survivors of Suicide Loss: A HEAL Report. J Clin Psychiatry. 2018 Mar/Apr;79(2):17m11592. doi: 10.4088/JCP.17m11592. PMID 29617064
- [Derived] Shear MK, Reynolds CF 3rd, Simon NM, Zisook S, Wang Y, Mauro C, Duan N, Lebowitz B, Skritskaya N. Optimizing Treatment of Complicated Grief: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Jul 1;73(7):685-94. doi: 10.1001/jamapsychiatry.2016.0892. PMID 27276373
- See also: Complicated Grief Research Group at University of Pittsburgh Medical Center — http://www.healstudy.org
- See also: Complicated Grief Program at Columbia University, New York — http://www.complicatedgrief.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Bereaved individuals age 18-95 were recruited between March 2010 and September 2014 using professional and public outreach, print, broadcast and internet media. Referrals were made by health care professionals, bereavement counselors and patients or family members.
Groups:
- Citalopram: Citalopram is an Selective Serotonin Reuptake Inhibitor (SSRI) medication. It is combined with grief-focused clinical management.
  Citalopram: 16 weeks of medication provided flexibly up to 40 mg/day. Medication is administered in a double-blind fashion.
- Placebo (Sugar Pill): Inactive medication. It is combined with grief-focused clinical management.
  Placebo: 16 weeks of daily inactive medication. It is administered in a double-blind fashion.
- CGT With Citalopram: The targeted psychotherapy for complicated grief combined with SSRI medication.
  Complicated Grief Treatment: Complicated Grief Treatment (CGT) is a targeted psychotherapy for complicated grief. The treatment integrates principles, strategies and techniques from interpersonal psychotherapy, trauma-focused cognitive behavioral treatment and motivational interviewing. Treatment includes 16 sessions provided within 20 weeks.
  Citalopram: 16 weeks of medication provided flexibly up to 40 mg/day. Medication is administered in a double-blind fashion.
- CGT With Placebo: The targeted psychotherapy for complicated grief combined with inactive medication.
  Complicated Grief Treatment: Complicated Grief Treatment (CGT) is a targeted psychotherapy for complicated grief. The treatment integrates principles, strategies and techniques from interpersonal psychotherapy, trauma-focused cognitive behavioral treatment and motivational interviewing. Treatment includes 16 sessions provided within 20 weeks.
  Placebo: 16 weeks of daily inactive medication. Medication is administered in a double-blind fashion.
Period: Overall Study
Arm/Group | Citalopram | Placebo (Sugar Pill) | CGT With Citalopram | CGT With Placebo
Started | 101 | 99 | 99 | 96
Completed Week 12 Assessment | 69 | 69 | 76 | 75
Completed (Week 20 assessment) | 73 | 61 | 76 | 76
Not Completed | 28 | 38 | 23 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Citalopram | Placebo (Sugar Pill) | CGT With Citalopram | CGT With Placebo | Total
Number analyzed (Participants) | 101 | 99 | 99 | 96 | 395
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (13.1) | 53.9 (13.8) | 52.1 (15.3) | 53.5 (16.0) | 53.0 (14.5)
Gender [Count of Participants; unit: Participants]
  Female | 82 | 69 | 78 | 79 | 308
  Male | 19 | 30 | 21 | 17 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 8 | 20 | 45
  Not Hispanic or Latino | 91 | 92 | 91 | 76 | 350
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  While | 85 | 80 | 81 | 79 | 325
  Black | 10 | 8 | 11 | 10 | 39
  Others | 6 | 11 | 7 | 7 | 31

OUTCOME MEASURES:

1. Primary Outcome: Responder Status Based on Complicated Grief Clinical Global Impression-Improvement (CGI-I) Scale
Description: Brief rating scale frequently used in clinical trials. For this study, version modified for complicated grief was be used. Response is defined as a score of 1(very much improved) or 2 (much improved) on the scale. The rating was done by an Independent Evaluator.
Time Frame: Weeks 12 and 20
Population: Response rates were compared under the intention-to-treat principle, including all randomized participants in a logistic regression with inverse probability weighting .
Measure: Number; unit: percentage of responders
Groups:
- Citalopram (CIT): Citalopram is an Selective Serotonin Reuptake Inhibitor (SSRI) medication. It is combined with grief-focused clinical management.
  Citalopram: 16 weeks of medication provided flexibly up to 40 mg/day. Medication is administered in a double-blind fashion.
- Placebo (PLA; Sugar Pill): Inactive medication. It is combined with grief-focused clinical management.
  Placebo (PLA): 16 weeks of daily inactive medication. It is administered in a double-blind fashion.
- Complicated Grief Treatment With Citalopram (CGT With CIT): The targeted psychotherapy for complicated grief combined with SSRI medication.
  Complicated Grief Treatment (CGT) is a targeted psychotherapy for complicated grief. The treatment integrates principles, strategies and techniques from interpersonal psychotherapy, trauma-focused cognitive behavioral treatment and motivational interviewing. Treatment includes 16 sessions provided within 20 weeks.
  Citalopram: 16 weeks of medication provided flexibly up to 40 mg/day. Medication is administered in a double-blind fashion.
- Complicated Grief Treatment With Placebo (CGT With PLA): The targeted psychotherapy for complicated grief combined with inactive medication.
  Complicated Grief Treatment (CGT) is a targeted psychotherapy for complicated grief. The treatment integrates principles, strategies and techniques from interpersonal psychotherapy, trauma-focused cognitive behavioral treatment and motivational interviewing. Treatment includes 16 sessions provided within 20 weeks.
  Placebo: 16 weeks of daily inactive medication. Medication is administered in a double-blind fashion.
Arm/Group | Citalopram (CIT) | Placebo (PLA; Sugar Pill) | Complicated Grief Treatment With Citalopram (CGT With CIT) | Complicated Grief Treatment With Placebo (CGT With PLA)
Number analyzed (Participants) | 101 | 99 | 99 | 96
percentage of responders | 46 | 38 | 84 | 83
Statistical Analysis 1: Comparison: Citalopram (CIT) vs Placebo (PLA; Sugar Pill); Our prespecified primary analysis was cross-sectional, comparing treatment response rates for CIT vs PLA at week 12 (aim 1), based on the intention-to-treat principle including all randomized participants. With 10% of 440 target enrollment lost to follow-up we had a power of 76-83% to detect predicted between-group difference in response (CGT with PLA, 40%; CGT with CIT, 60%; CIT 40%; and PLA 20%); Test type: Superiority or Other; p < 0.05, Regression, Logistic; Logistic regression with inverse probability weighting controlled for randomization stratification variables (site and baseline MDD) & race/ethnicity; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.82 to 1.81]
Statistical Analysis 2: Comparison: Complicated Grief Treatment With Citalopram (CGT With CIT) vs Complicated Grief Treatment With Placebo (CGT With PLA); Our prespecified primary analysis was cross-sectional, comparing treatment response rates for CIT with CGT vs PLA with CGT at week 20 (aim 2) based on the intention-to-treat principle including all randomized participants; Test type: Superiority or Other; p < 0.05, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.88 to 1.17]
Statistical Analysis 3: Comparison: Citalopram (CIT) vs Complicated Grief Treatment With Citalopram (CGT With CIT); Our prespecified primary analysis was cross-sectional, comparing treatment response rates for CIT with CGT vs CIT at week 20 (aim 3) based on the intention-to-treat principle including all randomized participants; Test type: Superiority or Other; p < 0.05, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.21, 95% CI 2-sided [1 to 1.46]

2. Secondary Outcome: Change From Baseline in Inventory of Complicated Grief (ICG)
Description: The 19-item self-report instrument assesses symptoms of complicated grief. Responses on individual items are added up to a total score, which can range from 0 to 76 with higher scores indicating more intense symptoms. This scale has been utilized previously in treatment studies of CG. Additional times points include weeks 4, 8, 12, 16, 20 and 40. For the pre-specified analyses we compared change in the ICG total score from baseline (calculated as baseline score minus week 12 score) for CIT vs PLA at week 12 (aim 1), based on the intention-to-treat principle including all randomized participants.
Time Frame: Baseline and week 12
Population: Prespecified secondary analyses of self-report ratings of CG symptoms (ICG) compared changes in scores using a weighted linear regression with inverse probability weighting to adjust for missing assessments.
Measure: Mean (Standard Deviation); unit: score change from baseline to wk12
Groups:
- Placebo (PLA; Sugar Pill): Inactive medication. It is combined with grief-focused clinical management.
  Placebo: 16 weeks of daily inactive medication. It is administered in a double-blind fashion.
Arm/Group | Citalopram (CIT) | Placebo (PLA; Sugar Pill)
Number analyzed (Participants) | 101 | 99
score change from baseline to wk12 | 18 (11) | 16 (12)
Statistical Analysis 1: Comparison: Citalopram (CIT) vs Placebo (PLA; Sugar Pill); Test type: Superiority or Other; p = 0.74, Regression, Linear — Pre-specified secondary analyses compared changes in ICG scores using a weighted linear regression, controlling for site, baseline MDD, & race/ethnicity, and with inverse probability weighting to adjust for missing assessments; Mean Difference (Final Values) = 0.67, Standard Error of Mean 2.04

3. Secondary Outcome: Change From Baseline in Inventory of Complicated Grief (ICG)
Description: The 19-item self-report instrument assesses symptoms of complicated grief. Responses on individual items are added up to a total score, which can range from 0 to 76 with higher scores indicating more intense symptoms. This scale has been utilized previously in treatment studies of CG. Additional times points include weeks 4, 8, 12, 16, 20 and 40. For the pre-specified analyses we compared change in the ICG total score from baseline (calculated as baseline score minus week 20 score) for CIT with CGT vs PLA with CGT (aim 2), and for CIT with CGT vs CIT (aim 3) based on the intention-to-treat principle including all randomized participants.
Time Frame: Baseline and week 20
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score change from baseline to wk20
Groups:
- Complicated Grief Treatment With Citalopram (CGT With CIT): The targeted psychotherapy for complicated grief combined with SSRI medication.
  Complicated Grief Treatment: Complicated Grief Treatment (CGT) is a targeted psychotherapy for complicated grief. The treatment integrates principles, strategies and techniques from interpersonal psychotherapy, trauma-focused cognitive behavioral treatment and motivational interviewing. Treatment includes 16 sessions provided within 20 weeks.
  Citalopram: 16 weeks of medication provided flexibly up to 40 mg/day. Medication is administered in a double-blind fashion.
- Complicated Grief Treatment With Placebo (CGT With PLA): The targeted psychotherapy for complicated grief combined with inactive medication.
  Complicated Grief Treatment: Complicated Grief Treatment (CGT) is a targeted psychotherapy for complicated grief. The treatment integrates principles, strategies and techniques from interpersonal psychotherapy, trauma-focused cognitive behavioral treatment and motivational interviewing. Treatment includes 16 sessions provided within 20 weeks.
  Placebo: 16 weeks of daily inactive medication. Medication is administered in a double-blind fashion.
Arm/Group | Citalopram (CIT) | Complicated Grief Treatment With Citalopram (CGT With CIT) | Complicated Grief Treatment With Placebo (CGT With PLA)
Number analyzed (Participants) | 101 | 99 | 96
score change from baseline to wk20 | 20 (12) | 25 (14) | 26 (12)
Statistical Analysis 1: Comparison: Complicated Grief Treatment With Citalopram (CGT With CIT) vs Complicated Grief Treatment With Placebo (CGT With PLA); Test type: Superiority or Other; p = .53, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.26, Standard Error of Mean 1.98
Statistical Analysis 2: Comparison: Citalopram (CIT) vs Complicated Grief Treatment With Citalopram (CGT With CIT); Test type: Superiority or Other; p < .001, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -7.37, Standard Error of Mean 2.08

4. Secondary Outcome: Change From Baseline in Work and Social Adjustment Scale (WSAS)
Description: The WSAS is a modification of a scale introduced by Hafner and Marks (1976), consisting of 0-8 point ratings of the extent to which symptoms interfere with five areas of daily functioning: work, home management, private leisure, social leisure, and family relationships. It is a well-validated, widely used self-report measure. Additional time points include weeks 4, 8, 12, 16, and 40. A total score calculated as a sum of all items (possible range 0-40) was used in the analyses with higher scores indicating more impairment. For the pre-specified analyses we compared change in the WSAS total score from baseline (calculated as baseline score minus week 12 score) for CIT vs PLA at week 12 (aim 1), based on the intention-to-treat principle including all randomized participants.
Time Frame: Baseline and week 12
Population: Prespecified secondary analyses of self-report ratings of grief-related functional impairment (WSAS) compared changes in scores using a weighted linear regression with inverse probability weighting to adjust for missing assessments.
Measure: Mean (Standard Deviation); unit: score change from baseline to wk12
Arm/Group | Citalopram (CIT) | Placebo (PLA; Sugar Pill)
Number analyzed (Participants) | 101 | 99
score change from baseline to wk12 | 10 (11) | 8 (10)
Statistical Analysis 1: Comparison: Citalopram (CIT) vs Placebo (PLA; Sugar Pill); Test type: Superiority or Other; p = .59, Regression, Linear — Pre-specified secondary analyses compared changes in WSAS scores using a weighted linear regression, controlling for site, baseline MDD, & race/ethnicity, and with inverse probability weighting to adjust for missing assessments; Mean Difference (Final Values) = -0.84, Standard Error of Mean 1.57

5. Secondary Outcome: Change From Baseline in Work and Social Adjustment Scale (WSAS)
Description: The WSAS is a modification of a scale introduced by Hafner and Marks (1976), consisting of 0-8 point ratings of the extent to which symptoms interfere with five areas of daily functioning: work, home management, private leisure, social leisure, and family relationships. It is a well-validated, widely used self-report measure. Additional time points include weeks 4, 8, 12, 16, and 40. A total score calculated as a sum of all items (possible range 0-40) was used in the analyses with higher scores indicating more impairment. For the pre-specified analyses we compared change in the WSAS total score from baseline (calculated as baseline score minus week 20 score) for CIT with CGT vs PLA with CGT (aim 2), and for CIT with CGT vs CIT (aim 3) based on the intention-to-treat principle including all randomized participants.
Time Frame: Baseline and week 20
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score change from baseline to wk20
Arm/Group | Citalopram (CIT) | Complicated Grief Treatment With Citalopram (CGT With CIT) | Complicated Grief Treatment With Placebo (CGT With PLA)
Number analyzed (Participants) | 101 | 99 | 96
score change from baseline to wk20 | 10 (12) | 14 (10) | 16 (11)
Statistical Analysis 1: Comparison: Complicated Grief Treatment With Citalopram (CGT With CIT) vs Complicated Grief Treatment With Placebo (CGT With PLA); Pre-specified secondary analyses compared changes in WSAS scores using a weighted linear regression, controlling for site, baseline MDD, & race/ethnicity, and with inverse probability weighting to adjust for missing assessments; Test type: Superiority or Other; p = .40, Regression, Linear; Mean Difference (Final Values) = 1.20, Standard Error of Mean 1.44
Statistical Analysis 2: Comparison: Citalopram (CIT) vs Complicated Grief Treatment With Citalopram (CGT With CIT); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = .005, Regression, Linear; Mean Difference (Final Values) = -4.13, Standard Error of Mean 1.46

ADVERSE EVENTS:
Time Frame: 5 years
Description: We observed no serious adverse medication effects. CGT therapists monitored participant response to emotionally activating procedures; no serious untoward responses were documented.
Arm/Group | Citalopram | Placebo (Sugar Pill) | CGT With Citalopram | CGT With Placebo
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/99 | 1/99 | 0/96
Other Adverse Events (participants affected / at risk) | 0/101 | 0/99 | 0/99 | 0/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram (N=101) | Placebo (Sugar Pill) (N=99) | CGT With Citalopram (N=99) | CGT With Placebo (N=96)
death by suicide (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Review by the study team and Institutional Review Board determined that this death was not related to the research

LIMITATIONS AND CAVEATS:
Two limitations of note: 1) FDA lowered the maximum safe dose of study medication (citalopram) after the study started; 2) our recruitment rate was 90% of target, while the assessment drop-out rate was over double what we expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No